CLINICAL TRIAL: NCT03446053
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dosing, Dose-Escalating Phase 1b Study to Evaluate the Safety, PK, PD and Immunogenicity of N-Rephasin® SAL200 After Continuous IV Infusion in Healthy Volunteers
Brief Title: A Study to Evaluate the Safety, PK, PD, Immunogenicity of N-Rephasin® SAL200 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intron Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITB-101_1b
Record Dates: First submitted 2018-02-04; First posted 2018-02-26 (Actual); Results first posted 2021-10-08 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-09

CONDITIONS: Healthy Volunteers; Anti-Bacterial Agents; Methicillin-Resistant Staphylococcus Aureus; Methicillin-Sensitive Staphylococcus Aureus Infection
Keywords: Methicillin-Resistant Staphylococcus Aureus; Methicillin-Sensitive Staphylococcus Aureus; N-Rephasin SAL200

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-Rephasin® SAL200 (Experimental): Forty subjects will be randomly assigned to receive either N-Rephasin® SAL200 injection or a placebo administered by a 60-min intravenous infusion. Within each group, 8 subjects (6 active and 2 placebo) will receive a single dose of 6 mg/kg, followed by multiple ascending dose of 3, 6, 9, and 12 mg/kg/day.
  Interventions: Biological: N-Rephasin® SAL200
- INT200-Placebo (Placebo Comparator): Saline
  Interventions: Other: INT200-Placebo

INTERVENTIONS:
Biological: N-Rephasin® SAL200 — continuous intravenous infusion over 60 minutes
  Arms: N-Rephasin® SAL200
Other: INT200-Placebo — Formulation buffer except active ingredient for continuous intravenous infusion over 60 minutes
  Arms: INT200-Placebo

SUMMARY:
To evaluate the safety, pharmacokinetics, pharmacodynamics and immunogenicity of N-Rephasin® SAL200 following single and multiple ascending doses in healthy male volunteers after continuous intravenous infusion over 60 minutes.

DETAILED DESCRIPTION:
* Forty subjects will be randomly assigned to receive either N-Rephasin® SAL200 injection or a placebo administered by a 60-min intravenous infusion. Within each group, 8 subjects (6 active and 2 placebo) will receive a single dose of 6 mg/kg, followed by multiple ascending dose of 3, 6, 9, and 12 mg/kg/day. The clinical trial will be performed in sequence from the lowest level, and the progress of the next dose level will be determined based on the safety results in the previous dose level.
* Examinations by interview, physical examinations, and screening tests such as clinical laboratory tests and allergenicity will be conducted in volunteers within 4 weeks (-28~-2d) from the previous day ot this clinical trial (-1d) to select subjects who are judged eligible for the study.
* Eligible subjects will be called in the afternoon (-1d) to examine the allergenicity in the clinical center of Seoul National Unviersity Hospital.
* Allergen-free subjects will be hospitalized on -1d and assigned with each subject number. All subjects are advised to fast from 10:00 p.m. overnight to the next morning, except drinking water. In the morning (09:00 a.m.) on 1d, subjects in each group will be given N-Rephasin® SAL200 injection or a placebo administered by a 60-min intravenous infusion, After that, the clinical trial will be conducted according to the designated schedule.
* All subjects receiving at least one dose will undergo a post-study visit test after a certain period of time. Immunogenicity testing will be performed until approximately 50 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged between 20 and 45 years at screening
* Those whose body weight is between 50kg and 90kg, and BMI is between 18.0 and 27.0
* Subjects who have fully understood this clinical trial via detailed explanation, are willing to voluntarily participate in this study, and agree to give written informed consent and to follow all of trial-related rules.

Exclusion Criteria:

* Those who have clinically significant liver, kidney, nervous system, endocrine system, respiratory system, hemato-oncology, cardiovascular system, mental diseases or past history.
* Those who have been diagnosed or suspected infectious disease within 30 days prior to the first dose of study medication
* Those who have history of hypersensitivity to drugs containing N-Rephasin® SAL200 or other drugs (aspirin and antibiotics)
* Those who have taken other drugs containing N-Rephasin® SAL200.
* Those who are antibody-positive to N-Rephasin® SAL200
* Those who have SBP <90mmHg or DBP <50mmHg (otherwise SBP > 150mmHg or DBP > 100mmHg) in vital signs, when measured after a 3-minute rest in sitting position.
* Those who have medical history of drug abuse or positive to urine drug screening
* Has taken any prescription drugs or herbal medicines within 14 days prior to first dose of study medication; otherwise, has taken over-the-counter drugs or vitamins within 7 days prior to the first dose of study medication (However, if other conditions are appropriate upon judgment of the investigator, the subject may participate in this study.)
* Those who has taken other study medications within 3 months prior to the study medication
* Those who have donated whole blood within 2 months prior to the first dose of study medication or apheresis within 1 month, or received blood transfusion within 1 months prior to the first dose of study medication
* Those who smoke cigarettes or are found to be nicotine metabolite-positive in urinalysis
* Those who cannot continuously abstain from drinking alcohol (exceeding 21 units/week, 1 unit = 10g of pure alcohol) or smoking cigarettes during hospitalization
* Those who are judged ineligible for the clinical study by the investigator due to other reasons, including the results of clinical laboratory tests
* Those who do not agree to use medically accepted contraceptive measures for 60 days after the first dose of study medication, or those who are unwilling to report the partner's pregnancy until 90 days after the first dose of study medication

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: In Jin Jang, M.D., Ph. D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Etienne J, Fleurette J, Ninet JF, Favet P, Gruer LD. Staphylococcal endocarditis after dental extraction. Lancet. 1986 Aug 30;2(8505):511-2. doi: 10.1016/s0140-6736(86)90377-6. No abstract available. PMID 2875256
- [Background] Kundsin RB. Documentation of airborne infection during surgery. Ann N Y Acad Sci. 1980;353:255-61. doi: 10.1111/j.1749-6632.1980.tb18928.x. No abstract available. PMID 6939390
- [Background] van Hal SJ, Jensen SO, Vaska VL, Espedido BA, Paterson DL, Gosbell IB. Predictors of mortality in Staphylococcus aureus Bacteremia. Clin Microbiol Rev. 2012 Apr;25(2):362-86. doi: 10.1128/CMR.05022-11. PMID 22491776
- [Derived] Wire MB, Jun SY, Jang IJ, Lee SH, Hwang JG, Huang DB. A Phase 1 Study To Evaluate Safety and Pharmacokinetics following Administration of Single and Multiple Doses of the Antistaphylococcal Lysin LSVT-1701 in Healthy Adult Subjects. Antimicrob Agents Chemother. 2022 Mar 15;66(3):e0184221. doi: 10.1128/AAC.01842-21. Epub 2022 Jan 10. PMID 35007129
- See also: Seung-Ho Han et al., Monitoring of Methicillin-Resistant Staphylococcus aureus in Nasal Swabs Obtained fron Dental Clinic Healthcare Providers and Medical Environments Nurses. Int J Oral Biology. 2010;35:7-12 — https://www.kci.go.kr/kciportal/ci/sereArticleSearch/ciSereArtiView.kci?sereArticleSearchBean.artiId=ART001432619
- See also: Eun Ja Park et al., Analysis of Economic Outcome of Methicillin-Resistant Staphylococcus aureus(MRSA) Bacteremia Using Retrospective Case-Control Study, Kor. J. Clin. Pharm 2007;17:59-64 — https://www.semanticscholar.org/paper/Analysis-of-Economic-Outcomes-of-Staphylococcus-Park-Chae/f848ff1bc9cf6e346dbbc24bd4b4bf669dd70b43
- See also: Hyuk Min Lee, Dong Eun Yong, Kyungwon Lee., Antimicrobial Resistance of Clinically Important Bacteria Isolated from 12 Hospitals in Korea in 2004 . Korean Journal of Clinical Microbiology 2005;8(1):66-73 — https://ir.ymlib.yonsei.ac.kr/handle/22282913/147505
- See also: Frency J, Brun Y, Bes M, Meugnier H, Grimont F, Grimon PAD, Newi C, Fleurette J. Staphylococcus lugdunensis sp. and Staphylococcus schleiferi sp. novel two species from human clinical specimens. Int Syst Bacteriol. 1998;38:168-172 — https://www.microbiologyresearch.org/content/journal/ijsem/10.1099/00207713-38-2-168

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was conducted in a single center (SEOUL NATIONAL UNIVERSITY HOSPITAL) from Feb. 2018 to Dec. 2018.
Pre-assignment Details: 59 subjects were screened and 33 subjects met inclusion criteria and were randomized to treatment.
Groups:
- Placebo, Single Dose Study: INT200-Placebo, single dose, IP administration: 1d 0h
- N-Rephasin® SAL200 6mg/kg (Single Dose): Sigle dose group N-Rephasin® SAL200 6mg/kg (single dose)
  Experimental: N-Rephasin® SAL200
  Active ingredient : SAL200 1ml (SAL-1 18 mg/mL) Manufacturer: BINEX Co., Ltd. (whole process contracted) Transparent and colorless vial filled with colorless clear liquid injection
  continuous intravenous infusion over 60 minutes
  Healthy Volunteers who were met eligibility criteria.
- Placebo , Multiple Dose Study: INT200-Placebo, multiple dose, IP administration: 1d 0h, 2d 0h, 2d 12h, 3d 0h, 3d 12h and 4d 0h
- N-Rephasin® SAL200 1.5 mg/kg (3mg/kg/d) , Multi Dose; N-Rephasin® SAL200 3mg/kg (6mg/kg/d), Multi Dose; N-Rephasin® SAL200 4.5mg/kg (9mg/kg/d), Multi Dose: multi dose study Experimental: N-Rephasin® SAL200
  Active ingredient : SAL200 1ml (SAL-1 18 mg/mL) Manufacturer: BINEX Co., Ltd. (whole process contracted) Transparent and colorless vial filled with colorless clear liquid injection
  continuous intravenous infusion over 60 minutes
  Healthy Volunteers who were met eligibility criteria.
Period: Overall Study
Arm/Group | Placebo, Single Dose Study | N-Rephasin® SAL200 6mg/kg (Single Dose) | Placebo , Multiple Dose Study | N-Rephasin® SAL200 1.5 mg/kg (3mg/kg/d) , Multi Dose | N-Rephasin® SAL200 3mg/kg (6mg/kg/d), Multi Dose | N-Rephasin® SAL200 4.5mg/kg (9mg/kg/d), Multi Dose
Started | 2 | 6 | 6 | 7 | 6 | 6
Randomized Set | 2 | 6 | 6 | 7 | 6 | 6
Safety Analysis Set | 2 | 6 | 6 | 6 | 6 | 6
PK/PD Analysis Set | 2 | 6 | 6 | 6 | 6 | 5
Completed | 2 | 5 | 6 | 6 | 6 | 5
Not Completed | 0 | 1 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- INT200-Placebo (Single Dose Study + Multi Dose Study): Saline
  INT200-Placebo: Formulation buffer except active ingredient for continuous intravenous infusion over 60 minutes
- N-Rephasin® SAL200 6mg/kg (Single Dose): Sigle dose N-Rephasin® SAL200 6mg/kg (single dose)
  Experimental: N-Rephasin® SAL200
  Active ingredient : SAL200 1ml (SAL-1 18 mg/mL) Manufacturer: BINEX Co., Ltd. (whole process contracted) Transparent and colorless vial filled with colorless clear liquid injection
  continuous intravenous infusion over 60 minutes
  Healthy Volunteers who were met eligibility criteria.
- N-Rephasin® SAL200 1.5 mg/kg (3mg/kg/d), Multi Dose; N-Rephasin® SAL200 3mg/kg (6mg/kg/d), Multi Dose; N-Rephasin® SAL200 4.5mg/kg (9mg/kg/d), Multi Dose: Multi dose Experimental: N-Rephasin® SAL200
  Active ingredient : SAL200 1ml (SAL-1 18 mg/mL) Manufacturer: BINEX Co., Ltd. (whole process contracted) Transparent and colorless vial filled with colorless clear liquid injection
  continuous intravenous infusion over 60 minutes
  Healthy Volunteers who were met eligibility criteria.
- Total: Total of all reporting groups
Arm/Group | INT200-Placebo (Single Dose Study + Multi Dose Study) | N-Rephasin® SAL200 6mg/kg (Single Dose) | N-Rephasin® SAL200 1.5 mg/kg (3mg/kg/d), Multi Dose | N-Rephasin® SAL200 3mg/kg (6mg/kg/d), Multi Dose | N-Rephasin® SAL200 4.5mg/kg (9mg/kg/d), Multi Dose | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 32
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 29.0 (5.6) | 28.5 (6.0) | 33.5 (6.2) | 31.3 (5.8) | 29.2 (4.9) | 30.2 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 6 | 6 | 6 | 6 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8 | 6 | 6 | 6 | 6 | 32
Weight [Mean (Standard Deviation); unit: kg] | 77.2 (8.8) | 73.1 (5.5) | 70.3 (9.1) | 74.2 (5.9) | 69.1 (8.7) | 73.0 (7.9)
Height [Mean (Standard Deviation); unit: cm] | 178.1 (6.2) | 175.0 (4.6) | 174.0 (3.6) | 174.5 (2.5) | 174.7 (4.9) | 175.4 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Evaluation
Description: Monitoring of adverse events (AEs) for Safety and Tolerability Evaluation
Time Frame: Up to 50D (±2D)
Measure: Count of Participants; unit: Participants
Groups:
- N-Rephasin® SAL200 (6mg/kg), Single Dose Study: SAL200 1 ml (SAL-1 18 mg/mL), 6 mg/kg, single dose, IP administration: 1d 0h
- N-Rephasin® SAL200 (1.5 mg/kg), Multiple Dose Study: SAL200 1 ml (SAL-1 18 mg/mL), 1.5 mg/kg (3 mg/kg/day), Multiple dose, IP administration: 1d 0h, 2d 0h, 2d 12h, 3d 0h, 3d 12h and 4d 0h
- N-Rephasin® SAL200 (3 mg/kg), Multiple Dose Study: SAL200 1 ml (SAL-1 18 mg/mL), 3 mg (6 mg/kg/day) , Multiple dose, IP administration: 1d 0h, 2d 0h, 2d 12h, 3d 0h, 3d 12h and 4d 0h
- N-Rephasin® SAL200 (4.5 mg/kg), Multiple Dose Study: SAL200 1 ml (SAL-1 18 mg/mL), 4.5 mg (9 mg/kg/day), Multiple dose, IP administration: 1d 0h, 2d 0h, 2d 12h, 3d 0h, 3d 12h and 4d 0h
Arm/Group | Placebo, Single Dose Study | N-Rephasin® SAL200 (6mg/kg), Single Dose Study | Placebo , Multiple Dose Study | N-Rephasin® SAL200 (1.5 mg/kg), Multiple Dose Study | N-Rephasin® SAL200 (3 mg/kg), Multiple Dose Study | N-Rephasin® SAL200 (4.5 mg/kg), Multiple Dose Study
Number analyzed (Participants) | 2 | 6 | 6 | 6 | 6 | 6
Participants
  No. of Subjects with TEAEs | 1 | 6 | 1 | 3 | 1 | 3
  No. of Subjects with Drug-Related TEAEs | 0 | 5 | 0 | 3 | 1 | 2
  No. of Subjects with Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0

2. Other Pre Specified Outcome: Pharmacokinetic Evaluation [Cmax (µg/mL)]
Description: Blood sampling for PK evaluation was performed at the following time points. Summary of PK parameters after single IV administration of N-Rephasin® SAL200.
Time Frame: Single administration: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours post-dose Multiple administration: the above timepoints and 25, 36, 48, 49, 60, 72, 72.25, 72.5, 72.75, 73, 73.5, 74, 75, 76, 77, 78, 80, 82, 84, 96 hours post-dose
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- N-Rephasin® SAL200 (6mg/kg): SAL200 1 ml (SAL-1 18 mg/mL), 6 mg/kg, single dose
- N-Rephasin® SAL200 (1.5 mg/kg): SAL200 1 ml (SAL-1 18 mg/mL), 1.5 mg/kg (3 mg/kg/day), single IV administration of N-Rephasin® SAL200
- N-Rephasin® SAL200 (3 mg/kg): SAL200 1 ml (SAL-1 18 mg/mL), 3 mg (6 mg/kg/day) , single IV administration
- N-Rephasin® SAL200 (4.5 mg/kg): SAL200 1 ml (SAL-1 18 mg/mL), 4.5 mg (9 mg/kg/day), single IV administration
Arm/Group | N-Rephasin® SAL200 (6mg/kg) | N-Rephasin® SAL200 (1.5 mg/kg) | N-Rephasin® SAL200 (3 mg/kg) | N-Rephasin® SAL200 (4.5 mg/kg)
Number analyzed (Participants) | 6 | 6 | 6 | 5
µg/mL | 21.4 (3.91) | 1.24 (0.509) | 4.93 (1.08) | 10.8 (1.53)

3. Other Pre Specified Outcome: Pharmacodynamic Evaluation
Description: Ex vivo antibacterial activity was assessed by bactericidal effects of the serum specimens collected from the trials were compared with calibration samples range of 0.05 to 1.0 μg/mL N-Rephasin®SAL200.
Time Frame: Up to 2hours
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- 6 mg/kg; 3 mg/kg; 4.5 mg/kg: single IV administration of N Rephasin® SAL200 IV administration.
- 1.5 mg/kg: after single IV administration of N Rephasin® SAL200 IV administration.
Arm/Group | 6 mg/kg | 1.5 mg/kg | 3 mg/kg | 4.5 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 5
μg/mL
  1.5h Mean concentration of bactericidal activity (μg/mL) | 0.38 (0.24) | 0.14 (0.20) | 0.22 (0.10) | 0.20 (0.00)
  2h Mean concentration of bactericidal activity (μg/mL) | 0.12 (0.07) | 0.02 (0.03) | 0.07 (0.07) | 0.08 (0.07)

4. Other Pre Specified Outcome: Immunogenicity Evaluation
Description: Anti-drug antibody titer was assessed.
Time Frame: Up to 50D (±2D)
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Single Dose Study + Multi Dose Study): INT200-Placebo (single dose study (2 participants) + multi dose study (6 participants) = total 8 participants)
- SAL200 N-Rephasin® SAL200 (6mg/kg) (Single Dose Study): SAL200 1 ml (SAL-1 18 mg/mL) , 6 mg/kg (Single dose study)
- SAL200 1.5 mg/kg (3 mg/kg/d) (Multi Dose Study): SAL200 1 ml (SAL-1 18 mg/mL), 1.5 mg/kg (3 mg/kg/day) (Multi dose study)
- SAL200 3 mg/kg (6 mg/kg/d) (Multi Dose Study): SAL200 1 ml (SAL-1 18 mg/mL), 3 mg (6 mg/kg/day) (Multi dose study)
- SAL200 4.5 mg/kg (9 mg/kg/d) (Multi Dose Study): SAL200 1 ml (SAL-1 18 mg/mL), 4.5 mg (9 mg/kg/day) (Multi dose study)
Arm/Group | Placebo (Single Dose Study + Multi Dose Study) | SAL200 N-Rephasin® SAL200 (6mg/kg) (Single Dose Study) | SAL200 1.5 mg/kg (3 mg/kg/d) (Multi Dose Study) | SAL200 3 mg/kg (6 mg/kg/d) (Multi Dose Study) | SAL200 4.5 mg/kg (9 mg/kg/d) (Multi Dose Study)
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 5
Participants
  ADA present at baseline | 0 | 0 | 0 | 0 | 0
  ADA negative at baseline | 8 | 6 | 6 | 6 | 5
  ADA positive post baseline (regardless of baseline) | 0 | 4 | 2 | 1 | 1
  ADA positive post baseline (baseline negative) | 0 | 4 | 2 | 1 | 1

5. Other Pre Specified Outcome: Pharmacokinetic Evaluation [AUClast, AUCinf (µg*h/mL)]
Description: as for outcome 2
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | N-Rephasin® SAL200 (6mg/kg) | N-Rephasin® SAL200 (1.5 mg/kg) | N-Rephasin® SAL200 (3 mg/kg) | N-Rephasin® SAL200 (4.5 mg/kg)
Number analyzed (Participants) | 6 | 6 | 6 | 5
µg*h/mL
  AUC last | 24.6 (7.04) | 1.10 (0.503) | 5.65 (1.33) | 11.3 (1.37)
  AUC inf | 24.8 (7.05) | 1.14 (0.519) | 5.70 (1.35) | 11.8 (1.15)

6. Other Pre Specified Outcome: Pharmacokinetic Evaluation [Tmax, T1/2, MRTinf (h)]
Description: as for outcome 2
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | N-Rephasin® SAL200 (6mg/kg) | N-Rephasin® SAL200 (1.5 mg/kg) | N-Rephasin® SAL200 (3 mg/kg) | N-Rephasin® SAL200 (4.5 mg/kg)
Number analyzed (Participants) | 6 | 6 | 6 | 5
h
  Tmax (h) | 1.00 (1.00) | 1.00 (1.00) | 1.00 (1.00) | 1.00 (1.00)
  T1/2 (h) | 3.38 (3.40) | 0.386 (0.0820) | 0.726 (0.214) | 1.16 (0.294)
  MRTinf (h) | 1.12 (0.314) | 0.656 (0.0760) | 0.782 (0.596) | 0.760 (0.0651)

7. Other Pre Specified Outcome: Pharmacokinetic Evaluation [Vd (L)]
Description: as for outcome 2
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: L
Arm/Group | N-Rephasin® SAL200 (6mg/kg) | N-Rephasin® SAL200 (1.5 mg/kg) | N-Rephasin® SAL200 (3 mg/kg) | N-Rephasin® SAL200 (4.5 mg/kg)
Number analyzed (Participants) | 6 | 6 | 6 | 5
L | 90.2 (89.5) | 55.6 (13.0) | 41.3 (9.82) | 46.4 (15.3)

8. Other Pre Specified Outcome: Pharmacokinetic Evaluation [CL (L/h)]
Description: as for outcome 2
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | N-Rephasin® SAL200 (6mg/kg) | N-Rephasin® SAL200 (1.5 mg/kg) | N-Rephasin® SAL200 (3 mg/kg) | N-Rephasin® SAL200 (4.5 mg/kg)
Number analyzed (Participants) | 6 | 6 | 6 | 5
L/h | 19.0 (5.63) | 107 (47.1) | 40.3 (5.89) | 27.4 (2.96)

ADVERSE EVENTS:
Time Frame: Up to 50 Days after randomization.
Groups:
- Placebo, Single Dose Study: INT200-Placebo (N=2),single dose study
- N-Rephasin® SAL200 (6mg/kg), Single Dose Study: N-Rephasin® SAL200 (6mg/kg), (N=6),single dose study
- Placebo , Multiple Dose Study: INT200-Placebo (N=6),multiple dose study
- N-Rephasin® SAL200 (1.5 mg/kg), Multiple Dose Study: N-Rephasin® SAL200 (1.5mg/kg), (N=6),multiple dose study
- N-Rephasin® SAL200 (3 mg/kg), Multiple Dose Study: N-Rephasin® SAL200 (3mg/kg), (N=6),multiple dose study
- N-Rephasin® SAL200 (4.5 mg/kg), Multiple Dose Study: N-Rephasin® SAL200 (4.5mg/kg), (N=6),multiple dose study
Arm/Group | Placebo, Single Dose Study | N-Rephasin® SAL200 (6mg/kg), Single Dose Study | Placebo , Multiple Dose Study | N-Rephasin® SAL200 (1.5 mg/kg), Multiple Dose Study | N-Rephasin® SAL200 (3 mg/kg), Multiple Dose Study | N-Rephasin® SAL200 (4.5 mg/kg), Multiple Dose Study
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/2 | 6/6 | 1/6 | 3/6 | 1/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo, Single Dose Study (N=2) | N-Rephasin® SAL200 (6mg/kg), Single Dose Study (N=6) | Placebo , Multiple Dose Study (N=6) | N-Rephasin® SAL200 (1.5 mg/kg), Multiple Dose Study (N=6) | N-Rephasin® SAL200 (3 mg/kg), Multiple Dose Study (N=6) | N-Rephasin® SAL200 (4.5 mg/kg), Multiple Dose Study (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — General disorders and administration site conditions
Pyrexia (General disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — General disorders and administration site conditions
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — General disorders and administration site conditions
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — General disorders and administration site conditions
Infusion site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — General disorders and administration site conditions
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) — General disorders and administration site conditions
Infusion site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — General disorders and administration site conditions
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — General disorders and administration site conditions
Ligament pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT03446053/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT03446053/SAP_001.pdf